CLINICAL TRIAL: NCT05121870
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Trial to Evaluate the Efficacy and Safety of Human Umbilical Cord-derived Mesenchymal Stem Cells Combined With Standard Therapy in Patients With Decompensated Cirrhosis
Brief Title: Treatment With Human Umbilical Cord-derived Mesenchymal Stem Cells for Decompensated Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other); LanZhou University (Other); Renmin Hospital of Wuhan University (Other); Chinese PLA General Hospital (Other); Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCRC-ID202105
Record Dates: First submitted 2021-10-17; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs) (Experimental): standard of care (SOC) plus UC-MSCs
  Interventions: Biological: UC-MSCs
- Placebo (Placebo Comparator): SOC plus placebo.
  Interventions: Biological: Saline containing 1% Human serum albumin（solution without UC-MSCs）

INTERVENTIONS:
Biological: UC-MSCs — 3 does of UC-MSCs(6.0×10E7cells per time) intravenously at week 0, week 4, week 8.
  Arms: Human Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs)
Biological: Saline containing 1% Human serum albumin（solution without UC-MSCs） — 3 does of placebo intravenously at week 0, week 4, week 8.
  Arms: Placebo

SUMMARY:
Decompensated cirrhosis has a high overall mortality rate. There is a large unmet need for safe and alternative therapeutic potions. This clinical trial is to inspect the efficiency and safety of mesenchymal stem cells (MSCs) therapy for decompensated cirrhosis.

DETAILED DESCRIPTION:
Decompensated cirrhosis has a high overall mortality rate. Liver transplantation is still the most effective treatment for decompensated cirrhosis. However, the shortage of matched liver sources, high costs, and rejection after liver transplantation restrict the development of liver transplantation.

Mesenchymal stem cells (MSC) are a kind of pluripotent stem cells belonging to mesoderm, which mainly exist in connective tissue and organ interstitium. At present, MSC can be isolated and prepared from bone marrow, fat, synovium, bone, muscle, lung, liver, pancreas and amniotic fluid and umbilical cord blood . Due to its wide range of sources and self-proliferation and differentiation ability, MSCs have therapeutic potential for many diseases, including acute and chronic liver diseases.

In recent years, our team has carried out a series of clinical trials using umbilical cord-derived MSCs to treat patients with end-stage liver disease, decompensated cirrhosis, primary biliary cholangitis, and status after liver transplantation and found that MSCs therapy can significantly improve patient liver function, reduce post-transplantation rejection, reduce complications, improve quality of life, and improve survival. Other investigators have also found in clinical trials with MSCs from different sources that treatment with MSCs can improve MELD scores or liver function levels to varying degrees. However, some studies have found no significant difference between the treatment group and the control group, and MSCs may differentiate into hepatic stellate cells and have the risk of promoting liver fibrosis, it is believed that MSCs do not favor the improvement of liver function in these studies. Therefore, the therapeutic effects of MSCs need to be further validated by larger multicenter randomized controlled clinical trials.

The investigators will do a prospective, double-blind, multicentre, randomised trial to assess treatment with three intravenous doses of MSCs compared with placebo. 240 decompensated cirrhosis patients will be recruited in China.120 patients will receive i.v. transfusion 3 times of MSCs (6.0×10E7 cells per time) and the standard of care as the treated group. In addition, the 120 patients will receive placebo and standard of care as control group.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. Aged 18 to 75 years (including 18 and 75 years), male or female;
3. Patients diagnosed with decompensated liver cirrhosis based on clinical findings, laboratory tests, imaging findings and/or representative pathological findings (decompensated liver cirrhosis is defined as the occurrence of at least one serious complication, including esophageal and gastric varices bleeding, hepatic encephalopathy, ascites, spontaneous bacterial peritonitis and other serious complications);
4. Child-Turcotte-Pugh (CTP) score 7 to 12 points.

Exclusion Criteria:

1. Appearance of active variceal bleeding, overt hepatic encephalopathy (HE), refractory ascites or hepatorenal syndrome within 1 month prior to screening visit.
2. Uncontrolled severe infection within 2 weeks of screening.
3. Hepatitis B virus (HBV) DNA ≥ detection limit at the time of screening.
4. Patients with hepatitis B virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HBV for less than 12 months.
5. Patients with hepatitis C virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HCV for less than 12 months.
6. Patients under treatment with corticosteroids for autoimmune hepatitis for less than 6 months.
7. Trans-jugular intrahepatic portosystemic shunts (TIPS) insertion within 6 months prior to study inclusion.
8. Active drinkers with alcohol-related decompensated cirrhosis are unwilling to stop alcohol abuse after inclusion.
9. Severe jaundice (serum total bilirubin level ≥ 170μmol/L); Significant renal insufficiency (serum creatinine ≥ 1.2 times upper normal limit); Severe electrolyte abnormality (serum sodium level < 125 mmol/L); Severe leukopenia (white blood cell count < 1 × 10E9/L).
10. Patients with biliary obstruction, hepatic vein, portal vein, splenic vein thrombosis and portal vein spongiosis.
11. Patients with surgical history such as splenic cut-off flow and portal body shunt.
12. Patients with confirmed or suspected malignancies.
13. Patients with a prior history of major organ transplantation or complicated with significant disease of heart, lung, kidney, blood, endocrine and other systems.
14. Drug abuse, drug dependence and patients who receive methadone treatment or with psychosis.
15. HIV seropositivity.
16. Those who have received blood transfusion or other blood products within 1 month prior to screening visit.
17. Pregnancy, lactation or with recent fertility plan.
18. Highly allergic or have a history of severe allergies.
19. Participants in other clinical trials within the last 3 months.
20. Any other clinical condition which the investigator considers would make the patient unsuitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Model for End-Stage Liver Disease (MELD) score from baseline to 24th week | at 24th week
  The Model for End-stage Liver Disease (MELD) is a scoring system that evaluates the liver function reserve and prognosis of patients with chronic liver disease by creatinine, international normalized ratio (INR), and bilirubin-conjugated cirrhosis etiology.
  The MELD score is calculated by the formula: R = 9.6 × ln (creatinine mg/dl) + 3.8 × ln (bilirubin mg/dl) + 11.2 × ln (INR) + 6.4 × etiology, and the results are taken as integers. ( 0 for cholestatic and alcoholic cirrhosis and 1 for other causes of cirrhosis such as viruses).

SECONDARY OUTCOMES:
Change in MELD score from baseline to 48 weeks | up to 48 weeks
Incidence of each complication associated with decompensated cirrhosis | up to 48 weeks
liver transplant-free survival | up to 48 weeks
Incidence of liver failure | up to 48 weeks
plasma albumin (ALB) | up to 48 weeks
total bilirubin (TBIL) | up to 48 weeks
serum cholinesterase (CHE) | up to 48 weeks
prothrombin activity (PA) | up to 48 weeks
Child-Turcotte-Pugh (CTP) score | up to 48 weeks
  Child-Turcotte-Pugh (CTP) score is a scoring system that evaluates the liver function.
EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D) | up to 48 weeks
ChronicLiver Disease Questionnaire (CLDQ) | up to 48 weeks
Incidence of liver cancer | up to 48 weeks
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | up to 48weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, PhD, Study Chair — Beijing 302 Hospital
Locations (5):
- China (5):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Hainan hospital of Chinese PLA General Hospital, Sanya, Hainan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Beijing 302 Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.